CLINICAL TRIAL: NCT05896917
Title: Do 3D Printed Foot Orthoses Reduce Self-reported Pain?-a Randomised Controlled Study
Brief Title: Comparison of 3D Printed Foot Orthoses With Prefabricated Foot Orthoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Dr. Abu Zeeshan Bari, Principal Investigator, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMR-PO-2023-421/8
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Flexible Flatfoot
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This group will receive 3D Printed Foot Orthoses
  Interventions: Device: 3D Printed Foot Orthosis
- Control (Active Comparator): This group will receive Prefabricated Foot Orthoses
  Interventions: Device: Prefabricated Foot Orthosis

INTERVENTIONS:
Device: 3D Printed Foot Orthosis — 3D printed foot orthoses designed and fabricated at the Taibah University
  Arms: Experimental
Device: Prefabricated Foot Orthosis — Generic foot orthoses available commercially
  Other Names: Insoles
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare the effects of 3D printed insoles versus prefabricated insoles in otherwise healthy subjects with flatfoot condition.

The main question it aims to answer is:

* If 3D printed insoles are better in terms of fit, weight, durability, comfort, and effectiveness compared to prefabricated insoles.
* If 3D printed insoles are better in terms of reducing pain compared to prefabricated insoles.

Participants will be divided in two groups. One group will receive 3D printed insoles and other group will wear prefabricated insoles for four weeks. After four weeks, researchers will record their feedback about their insoles which will help them to compare the two insoles.

DETAILED DESCRIPTION:
The purpose of this research is to compare the effects of 3D printed insoles versus prefabricated insoles in flatfoot subjects. This study will recruit healthy adult subjects with flexible flat feet but otherwise good physical and mental health. They will be divided into groups of an equal number of people. Prefabricated insoles will be given to one group, while 3D printed insoles will be given to the other. Subjective feedback will be collected at week zero, when the subjects will be given the insoles to wear, and again at the end of fourth week. Statistical analysis will be used to determine whether or not there is a significant difference in the responses of the two groups. The results will help us in identifying which insoles are better than the other in terms of parameters described above.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above
* Flatfoot symptoms such as foot/calf pain and fatigue after prolonged walking
* Foot postural index ranging from 6 to 12
* No neurological or physical disabilities

Exclusion Criteria:

* Below 18 years of age
* Inability to understand or answer questions
* Any lower limb surgery within the past two years
* Any lower limb injury within the past six months
* Any neurological disorder affecting gait

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Will be measured at Week 0
  The Visual Analog Scale is a validated tool for assessing pain. It involves a 10-centimeter line with the starting point at 0 centimeters representing no pain and the end point at 10 centimeters representing severe pain. Patients mark their pain level on the line, and the distance from the starting point provides a numerical measure of pain intensity.
Visual Analog Scale | Will be measured at Week 4
  The Visual Analog Scale is a validated tool for assessing pain. It involves a 10-centimeter line with the starting point at 0 centimeters representing no pain and the end point at 10 centimeters representing severe pain. Patients mark their pain level on the line, and the distance from the starting point provides a numerical measure of pain intensity.
Quebec User Evaluation of Satisfaction with Assistive Technology questionnaire. | Will be measured at 4th week
  The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) questionnaire is a tool designed to assess user satisfaction with assistive technology (AT) devices.
  A modified version of the QUEST questionnaire that will be used here consists of various items related to different aspects of assistive device use, such as device effectiveness, comfort, durability, weight, and dimensions. Respondents will be asked to rate each item on a scale, ranging from 1 (Not Satisfied at All) to 5 (Very Satisfied), indicating their level of satisfaction with each statement.

CONTACTS AND LOCATIONS:
Overall Officials: Abu Z Bari, PhD, Principal Investigator — Taibah University
Locations (1):
- Medical Rehabilitation Hospital, Madinah, Medina Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in this study
Supporting Information: Study Protocol
Time Frame: immediately following publication till after 2 years
Access Criteria: Access to data will be determined by Taibah University's CMRS ethical committee. Authorized individuals, including researchers and institutions, can access participant data for research and validation. Requests undergo review based on scientific merit, requester qualifications, data use, and compliance. Secure data transfer methods are employed to prioritize confidentiality.

REFERENCES:
- [Derived] Bari AZ, Ahmed N, Farhan M, Al-Shenqiti A, Zafar MS. Comparing Prefabricated and 3D-Printed Foot Orthoses for the Management of Flat Foot Condition: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Apr 1;104(4):298-304. doi: 10.1097/PHM.0000000000002585. Epub 2024 Jul 3. PMID 38958259